CLINICAL TRIAL: NCT02060825
Title: The Use of Optical Oximetry in Determining Gastrointestinal Complications After the Hybrid Procedure
Status: Terminated | Type: Observational
Why Stopped: Difficulty in downloading and saving data from the oximetry machine.
Sponsor: Aymen N Naguib (Other)
Responsible Party: Sponsor-Investigator, Aymen N Naguib, Director of Pediatric Cardiothoracic Anesthesia, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB12-00687
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Regional saturation monitor: Patients undergoing surgical repair of hypoplastic left heart syndrome.
  Interventions: Device: Regional saturation monitor

INTERVENTIONS:
Device: Regional saturation monitor
  Other Names: Casmed

SUMMARY:
This project is evaluating the validity of regional saturation monitoring in evaluating changes in the mesenteric perfusion. Regional saturation monitoring is a standard of care in many institutions, including NCH. Advances in the technology and recent approval of the use of CASMED devices for this purpose will allow us to use this technology more effectively. We aim to evaluate if there is a change in the mesenteric blood flow during the pre, intra and post operative period for the hybrid procedure and the balloon atrial septostomy procedure (BAS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of single ventricle and undergoing the hybrid procedure pathway.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgical repair of hypoplastic left heart syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Intestinal perfusion | Immediate post-op period (24 - 96 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States